CLINICAL TRIAL: NCT02617914
Title: Hemodynamic and Cardiac Effects of Individualized PEEP Titration Using Esophageal Pressure Measurements in ARDS Patients
Acronym: ENCODE
Status: Withdrawn | Type: Observational
Why Stopped: No approval from EC obtained. More details for study were required by EC.
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 15-122
Record Dates: First submitted 2015-11-23; First posted 2015-12-01 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Severe Acute Respiratory Distress Syndrome / Severe ARDS; Invasive Mechanical Ventilation; Individualized PEEP Treatment Strategy
Keywords: ARDS; PEEP; ECMO
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: individualized PEEP treatment, Invasive mechanical ventilation, ECMO,

SUMMARY:
The acute respiratory distress syndrome (ARDS) is common condition in critical ill patients affecting 7.2 people / 100,000 population / year and more than 7% of patients with invasive mechanical ventilation for more than 24 hours. ARDS carries a high hospital mortality of up to 48% and consumes large amounts of critical care resources. ARDS patients often present with severe hypoxemia that is refractory to conventional treatment and are thus evaluated for extracorporeal membrane oxygenation (ECMO). However, uncertainty regarding the appropriate indication for ECMO and clinical evidence for ECMO as a rescue treatment are still controversial. In 2012 Grasso and colleagues therefore presented a case series of influenza A (H1N1) ARDS patients describing the use of esophageal pressure measurements for individualized PEEP titration to achieve an end expiratory plateau pressure of the lung (PPLATL) of 25cm H2O. After performing the measurements in 14 patients, ventilator settings could be adjusted in half of these patients by increasing PEEP which resulted in an increase of oxygenation measures to an extend that criteria for extracorporeal support where no longer met and conventional treatment with invasive mechanical ventilation could be continued. However, uncertainty remains as to whether these results are generalizable to ARDS of any cause. In addition, increasing PEEP might impact on cardiac function and might therefore be associated with clinical important hemodynamic effects in these patients.

The investigators aim to evaluate hemodynamic changes in patients with severe ARDS in which an individualized PEEP treatment strategy can be employed. ARDS will be defined and stratified according to the Berlin ARDS definition. A naso-gastric probe capable of measuring esophageal pressure will be inserted directly after admission to the ICU as previously described. Invasive mechanical ventilation and oesophageal pressure measurements will be done using the GE Healthcare Carescape R860 ventilator. A pulmonary artery catheters (Edwards CCOcomb) will be inserted to evaluate the hemodynamic parameters of cardiac output, pulmonary artery pressures and left atrial pressures. Volumetric parameters will be measured using tanspulmonary thermodilution devices (Edwards EV1000). Cardiac function will be addressed in addition by the use of a predefined echocardiography protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Patients referred to our ICU for treatment of ARDS of any cause with a P/F ratio < 150 and indication for continued maximum critical care therapy
2. Male or female aged > 18 years
3. Written informed consent prior to study participation
4. The subject is willing and able to follow the procedures outlined in the protocol

Exclusion Criteria:

1. Patients admitted for primarily left ventricular or biventricular heart failure who are exclusively in need of cardiac and not pulmonary mechanical assist
2. Pregnant and lactating females
3. Patient has been committed to an institution by legal or regulatory order
4. Participation in a parallel interventional clinical trial
5. The subject received an investigational drug within 30 days prior to inclusion into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients referred to our ICU (Criitical Care Unit) for treatment of ARDS of any cause with a P/F ratio < 150 and indication for continued maximum critical care therapy. Patients of childbearing age with ARDS will be included.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic changes in parameters of cardiac output | Within the first 6 hours after ICU admission
Hemodynamic changes in parameters of pulmonary artery pressure | Within the first 6 hours after ICU admission
Hemodynamic changes in parameters of left atrial pressures | Within the first 6 hours after ICU admission
Hemodynamic changes in volumetric parameters | Within the first 6 hours after ICU admission

SECONDARY OUTCOMES:
ICU length of stay | Within 28 days after ICU admission
Time of ventilator | Within 28 days after ICU admission
Necessity of ECMO support | Within 28 days after ICU admission
Hospital length of stay | Within 28 days after ICU admission
28-day mortality | Within 28 days after ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kersten, MD, Principal Investigator — Department of Cardiology, Pneumology, Vascular Medicine and Critical Care (Medical Clinic I), University Hospital Aachen, Germany

REFERENCES:
- [Background] Villar J, Blanco J, Anon JM, Santos-Bouza A, Blanch L, Ambros A, Gandia F, Carriedo D, Mosteiro F, Basaldua S, Fernandez RL, Kacmarek RM; ALIEN Network. The ALIEN study: incidence and outcome of acute respiratory distress syndrome in the era of lung protective ventilation. Intensive Care Med. 2011 Dec;37(12):1932-41. doi: 10.1007/s00134-011-2380-4. Epub 2011 Oct 14. PMID 21997128
- [Background] Ferguson ND, Fan E, Camporota L, Antonelli M, Anzueto A, Beale R, Brochard L, Brower R, Esteban A, Gattinoni L, Rhodes A, Slutsky AS, Vincent JL, Rubenfeld GD, Thompson BT, Ranieri VM. The Berlin definition of ARDS: an expanded rationale, justification, and supplementary material. Intensive Care Med. 2012 Oct;38(10):1573-82. doi: 10.1007/s00134-012-2682-1. Epub 2012 Aug 25. PMID 22926653
- [Background] Roch A, Lepaul-Ercole R, Grisoli D, Bessereau J, Brissy O, Castanier M, Dizier S, Forel JM, Guervilly C, Gariboldi V, Collart F, Michelet P, Perrin G, Charrel R, Papazian L. Extracorporeal membrane oxygenation for severe influenza A (H1N1) acute respiratory distress syndrome: a prospective observational comparative study. Intensive Care Med. 2010 Nov;36(11):1899-905. doi: 10.1007/s00134-010-2021-3. Epub 2010 Aug 19. PMID 20721530
- [Background] Noah MA, Peek GJ, Finney SJ, Griffiths MJ, Harrison DA, Grieve R, Sadique MZ, Sekhon JS, McAuley DF, Firmin RK, Harvey C, Cordingley JJ, Price S, Vuylsteke A, Jenkins DP, Noble DW, Bloomfield R, Walsh TS, Perkins GD, Menon D, Taylor BL, Rowan KM. Referral to an extracorporeal membrane oxygenation center and mortality among patients with severe 2009 influenza A(H1N1). JAMA. 2011 Oct 19;306(15):1659-68. doi: 10.1001/jama.2011.1471. Epub 2011 Oct 5. PMID 21976615
- [Background] Hubmayr RD, Farmer JC. Should we "rescue" patients with 2009 influenza A(H1N1) and lung injury from conventional mechanical ventilation? Chest. 2010 Apr;137(4):745-7. doi: 10.1378/chest.09-2915. No abstract available. PMID 20371522
- [Background] Mitchell MD, Mikkelsen ME, Umscheid CA, Lee I, Fuchs BD, Halpern SD. A systematic review to inform institutional decisions about the use of extracorporeal membrane oxygenation during the H1N1 influenza pandemic. Crit Care Med. 2010 Jun;38(6):1398-404. doi: 10.1097/CCM.0b013e3181de45db. PMID 20400902
- [Background] Grasso S, Terragni P, Birocco A, Urbino R, Del Sorbo L, Filippini C, Mascia L, Pesenti A, Zangrillo A, Gattinoni L, Ranieri VM. ECMO criteria for influenza A (H1N1)-associated ARDS: role of transpulmonary pressure. Intensive Care Med. 2012 Mar;38(3):395-403. doi: 10.1007/s00134-012-2490-7. Epub 2012 Feb 10. PMID 22323077
- [Background] Akoumianaki E, Maggiore SM, Valenza F, Bellani G, Jubran A, Loring SH, Pelosi P, Talmor D, Grasso S, Chiumello D, Guerin C, Patroniti N, Ranieri VM, Gattinoni L, Nava S, Terragni PP, Pesenti A, Tobin M, Mancebo J, Brochard L; PLUG Working Group (Acute Respiratory Failure Section of the European Society of Intensive Care Medicine). The application of esophageal pressure measurement in patients with respiratory failure. Am J Respir Crit Care Med. 2014 Mar 1;189(5):520-31. doi: 10.1164/rccm.201312-2193CI. PMID 24467647
- [Background] Dalton HJ, MacLaren G. Extracorporeal membrane oxygenation in pandemic flu: insufficient evidence or worth the effort? Crit Care Med. 2010 Jun;38(6):1484-5. doi: 10.1097/CCM.0b013e3181e08fff. No abstract available. PMID 20502139